CLINICAL TRIAL: NCT04130932
Title: The Effect of Flooring on Office Workers' Health and Behaviors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brent A. Bauer, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Health Services Research
Other Study IDs: 19-006733
Record Dates: First submitted 2019-10-16; First posted 2019-10-18 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal flooring (No Intervention): standard office flooring
- Ergonomic flooring (Experimental): Ergonomically designed flooring
  Interventions: Other: Ergonomic flooring

INTERVENTIONS:
Other: Ergonomic flooring — Specially designed flooring system to optimize ergonomics of participants
  Arms: Ergonomic flooring

SUMMARY:
Researchers are trying to better understand how offices and workspaces influence people's performance, behavior and health during the course of weeks and over long periods of time.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Must be adults between the ages of 18 and 60
* Ability to relocate to the Well Living Lab for 9 consecutive weeks
* Full-time Mayo Clinic employees (35+ hours per week)
* Report working a sedentary job (e.g., sit for >= 50% of their work time).
* Have a working mobile phone that can receive text messages
* Must be present for 80% of the study (minimum of 4 days per week)

Exclusion Criteria:

* Individuals who are shift-workers
* Individuals diagnosed with vascular diseases (i.e., Raynaud's disease, peripheral artery disease, etc.)
* Individuals with diagnosed neurological and psychiatric disorders that may have physical limitations
* Drug (illegal or prescription narcotic), nicotine, or alcohol dependency
* Women who are lactating, pregnant or intend to become pregnant during the duration of the study
* Individuals who are taking medications (either prescribed or over-the-counter) which may affect comfort levels (e.g., opiate based medications)
* Working in occupation requiring standing/stepping >50% of work time
* Report < 1 year at current job
* Hospitalization from either a physical or mental disorder in the past six months
* History of cardiovascular, pulmonary, metabolic, neurological, or orthopedic limitations that would prohibit occupational physical activity (e.g., standing, stepping, etc.)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Sickness, absence, presenteeism | 9 weeks
  Work Limitations Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Brent Bauer, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials